CLINICAL TRIAL: NCT04152538
Title: Changes in Quadriceps Muscular Activity in Patients After Total Knee Arthroplasty Compared to Healty Subjects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, clinical research menager, Istituto Clinico Humanitas
Other Study IDs: CLF19/03
Record Dates: First submitted 2019-07-30; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Arthroplasty, Knee Replacement; Musculoskeletal Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy subjects: Healthy subjects matched with TKA patients
  Interventions: Other: not intervention but investigation
- TKA patients: age greater than 18 years old and a recent TKA.
  Interventions: Other: not intervention but investigation

INTERVENTIONS:
Other: not intervention but investigation — possible differences in quadriceps muscular activity

SUMMARY:
During Total Knee Arthroplasty (TKA), joint undergo considerable stress, which causes neuromuscular activation deficits of the quadriceps femoris muscle.The aim of the study is to investigate differences in quadriceps neuromuscular activity in the acute phase after surgery.

DETAILED DESCRIPTION:
During Total Knee Arthroplasty (TKA), joint undergo considerable stress, which causes neuromuscular activation deficits of the quadriceps femoris muscle. The current phenomenon depends on a complex mechanism called Arthrogenic Muscle Inhibition (AMI). AMI has been studied only in sub-acute and chronic phase after TKA due to the invasive procedures employed in order to evaluate it; However, clinical observation and experimental studies suggest presence of this phenomenon also in the first postoperative days. The aim of the study is to investigate differences in quadriceps neuromuscular activity, in acute phase.

The study is a prospective observational study.15 healthy subjects and 15 patients scheduled for TKA will be recruited. Patients will be asked to perform three isokinetic taks in the same standardized biomechanical context in order to evaluate changes in quadriceps neuromuscular activity after surgery as primary outcome. Secondly, correlation between primary aim and pain perceived by the patient will be investigated. Moreover, patient's functional ability will be assessed using the Timed Up and Go Test (TUG). Data will be recorded the day before TKA, at one and three days after surgery.

At the end of data acquisition, normality and homogeneity of demographic variables will be assessed. Differences in the outcome measures will be investigated with the t student test (or with the related non-parametric tests) and by means of the mixed models repeated measures ANOVA test. Linear regression will be applied to evaluate any correlation between outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age: over 18 years.
* subjects eligible for TKA.

Exclusion Criteria:

* QAB (quadriceps activation battery) < 6 the day before the operation
* neurological or musculoskeletal diseases (different from the causes that which led the patient to the TKA), which may interfere with the quadriceps muscle activation or with motor performance of the subject.
* Uncooperative subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample and hospitalized patients
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in quadriceps muscle activity | day before surgery, first postoperative day, third postoperative day for TKA group
  Surface EMG, RMS peak (mV)

SECONDARY OUTCOMES:
Change in pain perception | day before surgery, first postoperative day, third postoperative day for TKA group
  Numeric Rating Scale (NRS) 0-10. A value of 0 represents absence of pain, whereas a value of 10 represents maximum pain
Change in walking ability | day before surgery, thurd postoperative day for TKA group
  Timed Up and Go (TUG) evaluated in seconds,

CONTACTS AND LOCATIONS:
Locations (1):
- Roberto Gatti, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT04152538/Prot_SAP_000.pdf